CLINICAL TRIAL: NCT01471015
Title: Darbe Administration in Newborns Undergoing Cooling for Encephalopathy
Acronym: DANCE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Mariana Baserga, Principal Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 49096
Record Dates: First submitted 2011-11-02; First posted 2011-11-11 (Estimated); Results first posted 2015-05-22 (Estimated); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Hypoxic Ischemic Encephalopathy
Keywords: Hypoxic Ischemic Encephalopathy; Cooling Therapy; HIE
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High dose Darbepoetin alfa (Active Comparator): 10 mcg/kg/dose Darbe x2 doses, with the first dose within 12 hours of delivery and the second dose at 7 days
  Interventions: Drug: Darbepoetin alfa
- Low dose Darbepoetin alfa (Active Comparator): 2 mcg/kg/dose Darbe x2, with the first dose given within 12 hours of delivery and the second dose given at 7 days old.
  Interventions: Drug: Darbepoetin alfa
- Placebo (Placebo Comparator): Placebo given x2 doses, with the first given within 12 hours of delivery and the second given at 7 days old
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Darbepoetin alfa — 10 mcg/kg/dose x2, with the first dose given as IV within 12 hours of delivery and the second dose given as IV or SQ at 7 days old.
  Arms: High dose Darbepoetin alfa
Drug: Darbepoetin alfa — 2 mcg/kg/dose x2, with the first dose given IV within 12 hours of delivery and the second dose given IV or SQ at 7 days old.
  Arms: Low dose Darbepoetin alfa
Drug: Placebo — Placebo given x2, with the first dose given IV within 12 hours of delivery and the second dose given IV or SQ at 7 days old
  Arms: Placebo

SUMMARY:
Selective head cooling or whole body hypothermia has become the standard of care for neonatal hypoxia-ischemia encephalopathy (HIE). Despite early intervention death or major neurodevelopmental disability still occurs in nearly 50% of infants ≥ 36 weeks gestational age (GA) treated with cooling. No additional therapies have proven to be efficacious in further reducing brain injury and impairment for these high risk infants. Neuroprotective strategies aimed at improving early childhood outcomes are still needed. An important area of study includes therapies that may complement the neuroprotective effects of hypothermia and promote neuronal regeneration, recovery and neurovascular remodeling. Among these therapies, erythropoiesis stimulating agents (ESA) have been shown to provide neuroprotection, improving short and long-term neurologic outcome in brain injury and HIE in neonatal and adult animal models. Parallel with neuroprotective effects in experimental settings, recent small clinical studies suggest improved outcomes after ESA administration in patients with severe traumatic brain injury and HIE. ESA may work through several important mechanisms including reduced inflammation, limited oxidative stress, decreased apoptosis and white matter injury, as well as via pro-angiogenic and neurogenic properties.

Darbepoetin alfa (Darbe), a recombinant human erythropoietin (EPO)-derived molecule, has an extended circulating half life and comparable biological activity to EPO, including activation of the EPO receptor. The proposed study is a Phase I/II dose safety and pharmacokinetic trial of early Darbe administered concurrent with hypothermia in human newborn infants with moderate to severe birth asphyxia. The long-term objectives of the proposed research are to reduce mortality and to decrease the risk of long-term disabilities in infants with HIE who survive beyond the newborn period.

ELIGIBILITY:
Inclusion Criteria:

Infants will be eligible for the DANCE trial if they have a gestational age > 36 weeks by best obstetric estimate, are < 12 hours old and have evidence of moderate-severe acute perinatal HIE. Eligibility will also include criteria presently used in the NICU to initiate hypothermia:

1. < 6 hours after birth
2. History of an acute perinatal event (abruption, cord prolapsed, severe fetal heart rate abnormality)
3. Severe fetal or early (< 1 hour age) neonatal acidosis: arterial pH ≤ 7.0 or a base deficit ≥ 16m mEq/ L
4. If a blood gas is not available or a blood gas at <1 hour of age has a pH between 7.01 and 7.15, or a base deficit is between 10 and 15.9 mEq/L, additional criteria will be required:

   * acute perinatal event AND
   * either a 10-min Apgar score ≤ 5 or assisted ventilation initiated at birth and continued for at least 10 minutes.

Exclusion Criteria:

1. Major congenital and/or chromosomal abnormalities
2. Prenatal diagnosis of brain abnormality or hydrocephalus
3. Severe growth restriction (< 1800g)
4. Central venous hematocrit > 65%, platelet count > 600,000/dL, and/or neutropenia (ANC < 500 µL)
5. Maternal history of major vascular thrombosis or multiple fetal losses (> 3 spontaneous abortions)
6. ECMO
7. Infant judged critically ill and unlikely to benefit from neonatal intensive care by the attending neonatologist

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2012-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Baserga, MD, Principal Investigator — University of Utah
Locations (7):
- United States (7):
  - University of New Mexico, Albuquerque, New Mexico
  - Vanderbilt University School of Medicine, Nashville, Tennessee
  - McKay Dee Hospital- Intermountain Healthcare, Ogden, Utah
  - University of Utah, Salt Lake City, Utah
  - Primary Children's Hospital, Salt Lake City, Utah
  - Intermountain Medical Center, Sandy City, Utah
  - University of Washington, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Dose Darbepoetin Alfa | Low Dose Darbepoetin Alfa | Placebo
Started | 10 | 10 | 10
Completed | 10 | 9 | 9
Not Completed | 0 | 1 | 1
Not completed — Death | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Darbepoetin Alfa | Low Dose Darbepoetin Alfa | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Mean (Full Range); unit: days] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 6 | 15
  Male | 6 | 5 | 4 | 15
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Adverse Events.
Description: Potential adverse events such as (but not limited to) alterations in blood pressure, secondary infections, neutropenia, thrombotic/vascular events, hematologic events (platelets, Hct level, polycythemia), and hepatic/renal function that are outside of normal range for the study population.
  Complications associated with HIE or cooling therapy will not be considered an AE for this study. AEs reported to be associated with cooling include: bleeding/thrombosis, persistent pulmonary hypertension of the newborn (PPHN), skin changes, arrhythmia, and persistent acidosis.
Time Frame: 30 days or until hospital discharge
Measure: Number; unit: participants
Arm/Group | High Dose Darbepoetin Alfa | Low Dose Darbepoetin Alfa | Placebo
Number analyzed (Participants) | 10 | 10 | 10
participants | 7 | 7 | 8

2. Primary Outcome: The Pharmacokinetic Profile of Darbe After the First Dose During Cooling
Description: The pharmacokinetic profile of Darbe wil be determined using "population" pharmacokinetic sampling in which babies will be randomized to have blood drawn at different intervals. Serum levels will be drawn at 4,12, 18, 24, 36, 60, and 72 hours post initial dose. Area under the plasma concentration versus time curve (AUC) will be used.
Time Frame: For 72 hours after first dose
Measure: Median (Inter-Quartile Range); unit: AUC (h*mU/L)
Arm/Group | High Dose Darbepoetin Alfa | Low Dose Darbepoetin Alfa
Number analyzed (Participants) | 10 | 10
AUC (h*mU/L) | 180,866 [146,568 to 199,680] | 26,555 [20,049 to 35,029]
Statistical Analysis 1: Comparison: High Dose Darbepoetin Alfa vs Low Dose Darbepoetin Alfa; Test type: Superiority or Other; p = 0.006, Wilcoxon (Mann-Whitney)

3. Primary Outcome: The Pharmacokinetic Profile of Darbe After the Second Dose.
Description: The pharmacokinetic profile of Darbe will be determined using "population" pharmacokinetic sampling in which babies will be randomized to have blood drawn at different intervals. A second dose of Darbe will be given at 7 days of age, and serum drug levels will be obtained at 12, 18, 24, and 36 hours post second dose. Area under the plasma concentration versus time curve (AUC) will be used.
Time Frame: For 36 hours after second dose
Measure: Median (Inter-Quartile Range); unit: AUC (h*mU/L)
Arm/Group | High Dose Darbepoetin Alfa | Low Dose Darbepoetin Alfa
Number analyzed (Participants) | 10 | 10
AUC (h*mU/L) | 56233 [54915 to 71260] | 10790 [7043 to 13493]
Statistical Analysis 1: Comparison: High Dose Darbepoetin Alfa vs Low Dose Darbepoetin Alfa; Test type: Superiority or Other; p = 0.003, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | High Dose Darbepoetin Alfa | Low Dose Darbepoetin Alfa | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/10 | 1/10
Other Adverse Events (participants affected / at risk) | 7/10 | 7/10 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose Darbepoetin Alfa (N=10) | Low Dose Darbepoetin Alfa (N=10) | Placebo (N=10)
Death (General disorders) | 0 | 1 | 1 — Multi-organ failure due to Hypoxic-Ischemic Encephalopothy
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose Darbepoetin Alfa (N=10) | Low Dose Darbepoetin Alfa (N=10) | Placebo (N=10)
Hypotension (Cardiac disorders) | 4 | 4 | 4 — Defined as systolic blood pressure </= to 50 mmHg requiring inotrope support
Pulmonary Hypertension (Cardiac disorders) | 2 | 3 | 1
Altered Hepatic Function (Hepatobiliary disorders) | 2 | 1 | 1 — Defined as aspartate aminotransferase (AST) >200 IU/L or alanine aminotransferase (ALT) >100 IU/L
Altered Renal Function (Renal and urinary disorders) | 3 | 6 | 3 — Defined as urine output <0.5 mL/k/h for >24 hours or serum creatinine >1.5 mg/dL
Seizures (Nervous system disorders) | 3 | 2 | 0 — New onset seizures that appeared after the first dose of study drug

LIMITATIONS AND CAVEATS:
Due to the small number of participants, infrequent adverse events may not have been detected. There is a lack of long-term follow up to assess for long-term safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No